CLINICAL TRIAL: NCT01854008
Title: Improving Physical Activity in Patients With Severe Chronic Obstructive Pulmonary Disease With Urban Walking Circuits
Brief Title: Urban Walking Circuits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Eulogio Pleguezuelos, MD PhD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WALURB-01
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Severe Chronic Obstructive Pulmonary Disease
Keywords: Exercise, Physical activity, Rehabilitation, COPD.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rehabilitation program more the urban circuit (Experimental): One group, the urban circuit group (UCG), received a triptych that included urban walking circuits,the remaining patients formed the non circuit group (NCG).These circuits can be obtained on the website http://www.mataro.cat/web/portal/ca/salut/salut_publica/itineraris/index
  Interventions: Other: rehabilitation more the urban circuit
- rehabilitation program non circuit group . (Experimental): One group, the urban circuit group (UCG), received a triptych that included urban walking circuits,the remaining patients formed the non circuit group (NCG)
  Interventions: Other: rehabilitation program but not given urbane circuits

INTERVENTIONS:
Other: rehabilitation more the urban circuit — included in a standard rehabilitation program + the urban circuit. A total of 32 urban walking circuits were developed jointly with the town hall of Mataró(124,000 in habitants)and were included in a triptych called "A PEU, FEM SALUT! Itineraris urbans per Mataró" http://www.mataro.cat/web/portal/ca/salut/salut_publica/itineraris/index
  Arms: rehabilitation program more the urban circuit
Other: rehabilitation program but not given urbane circuits — Only rehabilitation program and general recommendations on physical activity and lifestyle . No urbans circuits.
  Arms: rehabilitation program non circuit group .

SUMMARY:
The aim of this study was to assess the effectiveness of the implementation of walking urban circuits in increasing the level of physical activity and exercise capacity in severe chronic obstructive pulmonary disease (COPD) patients after being enrolled in a pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* severe COPD (post-bronchodilator Forced expiratory volume in one second (FEV1)/ Forced vital capacity (FVC) <0.7 and FEV1 <50%) and stable disease defined as no exacerbation, hospital admission or change in treatment in the previous three months.

Exclusion Criteria:

* The exclusion criteria were: other significant respiratory disease (bronchiectasis, lung fibrosis, asthma, etc.), active smoking, severe cardiovascular, neurological, musculoskeletal and/or metabolic pathology that could interfere with the results, alcoholism (>80g/day) or severe malnutrition (BMI<19kg/m2).

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
walked in meters in the six minute walking test (6MWT) | Unlike walking meters of baseline and one year
  The 6MWT was standardized following international recommendations. Oxygen saturation and heart rate were recorded throughout the test using a pulsioximeter (Digit ® Finger Oximeter, Smiths Medical PM, USA). Dyspnea was evaluated using the modified Borg scale at the beginning and end of the test

CONTACTS AND LOCATIONS:
Locations (1):
- Eulogio Pleguezuelos, Mataró, Barcelona, Spain

REFERENCES:
- [Derived] Pleguezuelos E, Perez ME, Guirao L, Samitier B, Ortega P, Vila X, Solans M, Riera A, Moreno E, Meri A, Miravitlles M. Improving physical activity in patients with COPD with urban walking circuits. Respir Med. 2013 Dec;107(12):1948-56. doi: 10.1016/j.rmed.2013.07.008. Epub 2013 Jul 23. PMID 23890958
- See also: Related Info — http://www.csdm.cat